CLINICAL TRIAL: NCT01049516
Title: Prolonged Exposure for PTSD Among OIF/OEF Personnel: Massed vs. Spaced Trials
Brief Title: Prolonged Exposure for Post Traumatic Stress Disorder (PTSD) Among Operation Iraqi Freedom/Operation Enduring Freedom (OIF/OEF) Personnel
Acronym: STRONG STAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: The University of Texas Health Science Center at San Antonio (Other); U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PT074199P13; W81XWH-08-2-0111
Record Dates: First submitted 2010-01-12; First posted 2010-01-14 (Estimated); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Posttraumatic Stress Disorders; Combat Disorders
Keywords: Military; Combat; Psychological Treatment; Psychotherapy; Trauma; Posttraumatic Stress; Posttraumatic Stress Disorder; PTSD; Prolonged Exposure; Exposure therapy; Behavior Therapy; Cognitive Behavior Therapy; Post-Traumatic Stress Disorders; Stress Disorders, Post-traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Combat Disorders; Wounds and Injuries | interventions — Waiting Lists

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Minimal Contact Control (Other)
  Interventions: Behavioral: Minimal Contact Control
- PE-Massed (Experimental)
  Interventions: Behavioral: Prolonged Exposure Therapy - Massed
- PE-Spaced (Active Comparator)
  Interventions: Behavioral: Prolonged Exposure Therapy - Spaced
- Present-Centered Therapy (PCT) (Active Comparator)
  Interventions: Behavioral: Present-Centered Therapy

INTERVENTIONS:
Behavioral: Prolonged Exposure Therapy - Massed — 10 75-90 minute psychotherapy sessions, focused on gradually confronting distressing trauma-related memories and reminders. Sessions occur 5 days/week for two weeks.
  Other Names: Massed-PE
  Arms: PE-Massed
Behavioral: Prolonged Exposure Therapy - Spaced — 10 75-90 minute psychotherapy sessions, focused on gradually confronting distressing trauma-related memories and reminders. Sessions 1-3 occur in the first two weeks, Sessions 4-5 occur in Weeks 3-4, and Sessions 6-10 occur in Weeks 5-10.
  Other Names: Spaced-PE
  Arms: PE-Spaced
Behavioral: Minimal Contact Control — Participants receive minimal contact for 4 weeks after randomization and thereafter are offered PE-Spaced or PE-Massed, according to their preference. Participants receive 10-15 minute phone calls once per week by the study therapist or independent evaluator in order to monitor their status and to provide support as needed.
  Other Names: Wait List
  Arms: Minimal Contact Control
Behavioral: Present-Centered Therapy — 10 75-90 minute psychotherapy sessions, focused on identifying and solving day-to-day problems as they are brought up by the participants
  Arms: Present-Centered Therapy (PCT)

SUMMARY:
The purpose of this study is 1) to evaluate whether massing 10 PE sessions in 2 weeks (massed trials; M-PE) is more efficacious than Minimal Contact control (MCC); 2) whether the massed sessions format retains the efficacy of treatment compared to 10 PE sessions spaced over 8 weeks (spaced trials; S-PE), and 3) to evaluate for the first time the efficacy of the 10 PE sessions delivered in 8 weeks in an active duty population by comparing it to an active comparison condition, Present-Centered Therapy (PCT).

DETAILED DESCRIPTION:
The purpose of this study is to improve the efficiency of treatment for post-traumatic stress disorder (PTSD) with prolonged exposure (PE), an efficacious treatment for PTSD typically administered in once- or twice-weekly sessions. We will evaluate whether massing 10 PE sessions in 2 weeks (massed trials; M-PE) is more efficacious than Minimal Contact control (MCC); 2) whether the massed sessions format retains the efficacy of treatment compared to 10 PE sessions spaced over 8 weeks (spaced trials; S-PE), and 3) will evaluate for the first time the efficacy of the 10 PE sessions delivered in 8 weeks in an active duty population by comparing it to an active comparison condition, Present-Centered Therapy (PCT). Randomization was initially set at 3:11:11:11 for MCC:M-PE:S-PE:PCT. Due to the urgent need for data to inform military clinical practice, enrollment in MCC was accelerated by changing the ratio to 1:1:1:1 in order to report the comparison between M-PE and MCC. When 30 participants were enrolled in MCC, randomization resumed to approximately 3:11:11:11. Prolonged Exposure (PE; Foa, Hembree, & Rothbaum, 2007; Foa & Rothbaum, 1998) was developed by the PI, Edna Foa, and colleagues in the Center for the Treatment & Study of Anxiety (CTSA), University of Pennsylvania. It has been found quite efficacious in reducing PTSD and related psychopathology with various types of trauma in PTSD centers around the world. Furthermore, PE has been identified in the joint VA-Department of Defense Clinical Practice Guideline for PTSD (VA-DoD Clinical Practice Guideline Working Group, 2003) as "strongly recommended" for use with veterans with PTSD, based on the strong empirical support for PE.

This study is part of the South Texas Research Organizational Network Guiding Studies on Trauma and Resilience (STRONG STAR) (Consortium Director: Alan L. Peterson, Ph.D., ABPP, Professor, Behavioral Wellness Center for Clinical Trials, Department of Psychiatry-Mail Code 7792, University of Texas Health Science Center at San Antonio (UTHSCSA), 7703 Floyd Curl Drive, San Antonio, TX 78229-3900). Dr. Edna Foa is the overall PI of the study, and the on-site PI is COL Jeffrey Yarvis, Ph.D.,Chief, Soldier Behavioral Health/Outpatient Psychiatry, Carl R. Darnall Army Medical Center, 36000 Darnall Loop, Fort Hood, TX, 76544. The study will be conducted at Fort Hood, Texas.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female active-duty OIF/OEF military personnel and recently separated OIF/OEF veterans ages 18-65 seeking treatment for PTSD
* Diagnosis of PTSD determined by a clinician-administered Posttraumatic Stress Scale (PSS-I).

Exclusion Criteria:

* Current bipolar disorder or other psychotic disorder (as determined by the evaluator conducting the patient interview and medical record review)
* Current alcohol dependence (as determined by the AUDIT)
* Evidence of a moderate or severe traumatic brain injury (as determined by the inability to comprehend the baseline screening questionnaires)
* Current suicidal ideation severe enough to warrant immediate attention (as determined by the Scale for Suicidal Ideation)
* Other psychiatric disorders severe enough to warrant designation as the primary disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2010-11; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Change in PTSD Symptom Scale, Interview Version (PSS-I) following treatment | Baseline to 6-month follow-up (approximately 34 weeks for Spaced PE and PCT, 26 weeks for Massed PE
  Affect of treatment on this measure of PTSD symptomology

SECONDARY OUTCOMES:
PTSD Checklist-Stressor-specific version (PCL-S) | Baseline to Post-treatment (approximately 10 weeks for Spaced PE and PCT, 2 weeks for Massed PE)
  Affect of treatment on a PTSD Assessment of stress
PTSD Checklist-Stressor-specific version (PCL-S) | Post-treatment to 2-week follow-up
  Changes in PTSD stress symptomology upon commencement of treatment
PTSD Checklist-Stressor-specific version (PCL-S) | 2-week follow-up to 12-week follow-up
  Changes in PTSD stress symptomology upon commencement of treatment
PTSD Checklist-Stressor-specific version (PCL-S) | 12-week follow-up to 6-month follow-up
  Changes in PTSD stress symptomology upon commencement of treatment
Changes in PTSD diagnosis using PTSD Symptom Scale, Interview Version (PSS-I) over course of treatment | Baseline to Post-treatment (approximately 10 weeks for Spaced PE and PCT, 2 weeks for Massed PE)
  PTSD Assessment
Changes in PTSD diagnosis using PTSD Symptom Scale, Interview Version (PSS-I) following treatment | Post-treatment to 2-week follow-up
  PTSD Assessment
Changes in PTSD diagnosis using PTSD Symptom Scale, Interview Version (PSS-I) following treatment | 2-week follow-up to 12-week follow-up
  PTSD Assessment
Changes in PTSD diagnosis using PTSD Symptom Scale, Interview Version (PSS-I) following treatment | 12-week follow-up to 6-month follow-up
  PTSD Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Edna B. Foa, Ph.D., Principal Investigator — Center for the Treatment and Study of Anxiety, University of Pennsylvania; Elna Yadin, Ph.D., Study Director — Center for the Treatment and Study of Anxiety, University of Pennsylvania
Locations (3):
- United States (3):
  - Center for the Treatment and Study of Anxiety, University of Pennsylvania, Philadelphia, Pennsylvania
  - Carl R. Darnall Army Medical Center, Killeen, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

REFERENCES:
- [Derived] Taylor DJ, Pruiksma KE, Hale W, McLean CP, Zandberg LJ, Brown L, Mintz J, Young-McCaughan S, Peterson AL, Yarvis JS, Dondanville KA, Litz BT, Roache J, Foa EB. Sleep problems in active duty military personnel seeking treatment for posttraumatic stress disorder: presence, change, and impact on outcomes. Sleep. 2020 Oct 13;43(10):zsaa065. doi: 10.1093/sleep/zsaa065. PMID 32246153
- [Derived] Brown LA, Zang Y, Benhamou K, Taylor DJ, Bryan CJ, Yarvis JS, Dondanville KA, Litz BT, Mintz J, Roache JD, Pruiksma KE, Fina BA, Young-McCaughan S, Peterson AL, Foa EB; STRONG STAR Consortium. Mediation of suicide ideation in prolonged exposure therapy for posttraumatic stress disorder. Behav Res Ther. 2019 Aug;119:103409. doi: 10.1016/j.brat.2019.103409. Epub 2019 May 23. PMID 31176888
- [Derived] Foa EB, McLean CP, Zang Y, Rosenfield D, Yadin E, Yarvis JS, Mintz J, Young-McCaughan S, Borah EV, Dondanville KA, Fina BA, Hall-Clark BN, Lichner T, Litz BT, Roache J, Wright EC, Peterson AL; STRONG STAR Consortium. Effect of Prolonged Exposure Therapy Delivered Over 2 Weeks vs 8 Weeks vs Present-Centered Therapy on PTSD Symptom Severity in Military Personnel: A Randomized Clinical Trial. JAMA. 2018 Jan 23;319(4):354-364. doi: 10.1001/jama.2017.21242. PMID 29362795
- See also: Link to Strong Star research consortium — https://delta.uthscsa.edu/strongstar/